CLINICAL TRIAL: NCT03609632
Title: Exploring Beta Cell Function in Individuals With Postbariatric Postprandial
Brief Title: Understanding Hypoglycaemia After Bariatric Surgery
Acronym: HYPOBAR1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Erasmus Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HYPOBAR1
Record Dates: First submitted 2018-07-25; First posted 2018-08-01 (Actual); Last update posted 2018-12-04 (Actual); Status verified 2018-12

CONDITIONS: Bariatric Surgery
Keywords: Roux-en-Y gastric bypass (RYGB); Hypoglycaemia; Insulin; Glucose; Incretins; Stable isotope
MeSH Terms: conditions — Hypoglycemia; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OGTT with 13C-labelled leucine (Experimental): Intake of 75g of glucose with 1g of 13C leucine pre-feeding
  Interventions: Other: Dietary Supplement: Glucose

INTERVENTIONS:
Other: Dietary Supplement: Glucose — Intake of 75g of glucose with 1g of 13C leucine pre-feeding

SUMMARY:
Postprandial hyperinsulinaemic hypoglycaemia is an increasingly recognized adverse side effect of bariatric surgery. Affected individuals experience low glucose levels 1-3 hours after intake of meals, accompanied by symptoms such as drowsiness, sweating, hunger and palpitations. Hypoglycaemia can be serious and have potential dangerous health impact (e.g. road accident or fall due to loss of consciousness). The pathophysiology is incompletely understood and more research is needed in search of preventive and therapeutic strategies.

DETAILED DESCRIPTION:
Obesity is a major global health concern that is associated with significant disability and mortality. Worldwide, the prevalence of obesity has doubled since 1980, affecting 13% of the global population. Bariatric surgery has been shown to be the most effective and durable treatment of severe obesity and leads to significant improvement of obesity-related comorbidity. However, postprandial hyperinsulinaemic hypoglycaemia (PHH) after bariatric surgery is a metabolic complication that is increasingly being recognized. Prevalence rates of up to 72% have been reported. PHH may have serious implications for affected patients, including negative effects on morbidity, mortality as well as quality of life. The pathophysiology of PPH is incompletely understood and suggests decreased adaptation of beta cell function to increased insulin sensitivity. The latter has been postulated to be largely secondary due to external factors outside the beta cells as a result of anatomical and hormonal changes after Roux-en-Y gastric bypass (RYGB). However, the intrinsic mechanistic effects of altered beta-cell function after RYGB in vivo are unknown and more exploration could lead to a better understanding of PHH pathogenesis and help identify targets for possible interventions. Previous studies performed enhanced beta cell analysis by following insulin synthesis in real-time based on stable isotope labelling of C-peptide during an oral glucose tolerance test (OGTT) in cohorts with normal and diabetic glucose tolerance. Applying the same methodological approach, albeit in a different target population (PPH after bariatric surgery), the present study seeks to explore whether or not the insulin hypersecretion can be explained by an increase in insulin synthesis, and secondly, whether potentially increased insulin synthesis can be related to other glucoregulatory hormones and measures of insulin sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Gastric bypass (RYGB) surgery performed ≥ 6 months ago
* Confirmed postprandial hypoglycaemia (continuous glucose monitoring or plasma glucose), with at least 2 episodes of Whipple's triad (symptoms, capillary of interstitial glucose ≤3.1mmol/L, symptom resolution by carbohydrate intake) ≤3 months ago
* Normal glucose control at recruitment and absence of (pre)diabetes before bariatric surgery
* Capacity to give informed consent

Exclusion Criteria:

* Fasting hypoglycaemia suggesting hyperinsulinism of different aetiology
* Use of medication that influence glucose metabolism
* Bariatric procedures other than RYGB
* Physical or psychological disease likely to interfere with the normal conduct of the study and interpretation of the study results as judged by the investigator
* Moderate to severe chronic kidney disease
* Pregnancy or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-09-20 (Actual); Primary Completion 2018-11-02 (Actual); Study Completion 2018-11-02 (Actual)

PRIMARY OUTCOMES:
Fractional synthesis rate of de novo C-peptide synthesis (%/hr) | 4.5 hours
  Calculated

SECONDARY OUTCOMES:
C-peptide levels in blood | 4.5 hours
  Measured
Insulin levels in blood | 4.5 hours
  Measured
Glucagon levels in blood | 4.5 hours
  Measured
Incretin levels in blood | 4.5 hours
  Measured
Insulin sensitivity | 4.5 hours
  Calculated
Beta cell responsivity | 4.5 hours
  Calculated
Hepatic insulin extraction | 4.5 hours
  Calculated
C-peptide levels in urine | 4.5 hours
  Measured
C-peptide enrichment | 4.5 hours
  calculated

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Stettler, MD, Principal Investigator — Inselspital, Bern University Hospital, University of Bern
Locations (1):
- Division of Endocrinology, Diabetes and Clinical Nutrition, Bern University Hospital, Bern, Switzerland